CLINICAL TRIAL: NCT02827396
Title: A Mixed Methods Study to Design and Test Effectiveness of a Psycho-social Training Intervention on Psychological Health of Parents for Intellectually Disabled Children in Malawi
Brief Title: Effectiveness of a Training Intervention on Mental Health of Parents for Intellectually Disabled Children in Malawi
Acronym: PSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St John of God, Malawi (Other)
Responsible Party: Principal Investigator, Charles Masulani Mwale, Director, St John of God, Malawi
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SJOG594
Record Dates: First submitted 2016-05-17; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Depression; Learning Disability
Keywords: Disability; children; parents; depression; knowledge; psychosocial intervention
MeSH Terms: conditions — Depression; Learning Disabilities | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psycho-social intervention (Experimental): Experimental group: The intervention group will get Psycho social Training Intervention which will be developed during the third phase of the study.
  Interventions: Behavioral: Psychosocial intervention
- TAU intervention (No Intervention): Wait-list (controlled) group: The waiting list (control) group will continue getting the general health education (TAU) that is done at disability clinics in the existing sites.

INTERVENTIONS:
Behavioral: Psychosocial intervention — This training is aimed at Mothers/Fathers/Caregivers/Grandparents of children with intellectual disabilities.
  Individual (for severe mental health problems) or group counseling for similar psychological issues should be a vital ingredient of this program. The package runs for 40 hours. It will run for five days continuously. It's important to promote participatory rather than deductive approach allow a lot of time for questions and discussions.
  Arms: Psycho-social intervention

SUMMARY:
Background: It is asserted that 85% of disabled children live in resource poor countries with few available disability services. Measurements have shown an increase in disability prevalence from 2% to 4% over the past three decades in Malawi. A recent prevalence study in Mzuzu city, found 19.7% disability prevalence with associated social and psychological burden of care; marriage disruptions and divorces among parents of disabled children due to stigma and cultural misconceptions about disability.

Studies have shown a link between parenting children with intellectual disabilities and parental psychological health problems and overall Quality of life. However, with interventions, these negative impacts are not as severe as once thought.

Research Objectives: This study aims to design a Malawi specific Psychosocial Training Intervention for parents with intellectually disabled children and assess the impact of the Intervention in reducing psychological distress among these parents in Malawi.

Methodology: This study will use mixed methods design. It will employ an explanatory sequential design, where by qualitative data collection and analysis builds to quantitative data collection and analysis; and final interpretation.

The study will be conducted within catchment areas of two disability organisations that are operating in Mzuzu and Lilongwe.

On sample size for the quantitative part, calculation using 5% level of statistical significance, power of 90% and effect size of 0.4 [effect size found in recent meta-analysis for similar intervention, gives 81 participants in each arm of the intervention. Questionnaire with social-demographic data in section one; and "Self-Reported Questionnaire will be administered at baseline, 6 & 12 months follow-up. Quantitative data will be coded on a computer, cleaned and analyzed using STATA. Mann-Whitney test will be used to measure the impact of the intervention. Qualitative data will be analysed using content analysis with the help of Nvivo.

All ethical consideration will be followed to ensure that subjects are treated with respect; allow for their right to refuse participation in the study; and conducting interviews in privacy.

Dissemination: Findings will be disseminated through Continous profesional development (CPD) sessions at the two clinic sites; Research Dissemination Conferences in Malawi and Sub-region; and three manuscripts submission for publication in peer reviewed journals.

DETAILED DESCRIPTION:
Background Information and Introduction:

It is argued that 85% of children with disability live in resource poor countries where there are few available disability services. A majority of these children, including their carers, suffer the double burden of disability and its associated stigmatization, leading to a marginalized life.

There has been an increase in disability prevalence in Malawi over the past three decades A 1983 National Statistical Office Survey of Handicapped Persons in Malawi, using head count and snowball sampling placed the rate of disability in the population at 2.9% and 10 years later it was estimated at 2%. However in a recent prevalence study in Mzuzu city, it was found that 154 out of the 780 children sampled (aged 0-18 years) have at least some kind of disability according to the Ten Question Questionnaire (a screening tool for disability in low income settings comprising five questions on cognitive development; two questions on motor development; and one question each regarding vision, hearing and seizures), representing 19.7% prevalence. The low prevalence in the earlier surveys may not have addressed multiple disabilities unlike in this study where a variety of disabilities including physical, intellectual and self-care were studied. In Mzuzu a significant burden of care was found among guardians of these children. Much of this related to stigma and cultural misconceptions about disability and its causes. Physical, social and psychological burdens were reported leading to children being locked up for fear of carrying heavy weight on the back as well as stigma; marriage disruptions and divorces between carers ; and general distress as a result of having a disabled child.

It is also clear therefore that in addition to the high burden of disease from childhood disability, mental health problems (in particular - depression) in carers only add to this burden of disease. To add on the issue of disability, asserts that depressive disorders are the leading causes of years lost due to disability in 2004.

There is no cure for most disabilities, including intellectual disabilities, but psycho-social interventions can help parents and carers of children with intellectual disabilities. Traditionally, researchers have believed that parenting these children has negative impacts on carers. These include increased psychological and physical health problems for carers; and physical, social, and financial distress to the whole family. This impact most on parents, as they are virtually the only constant carers; leading often to increased divorce rates. Recent studies from high income settings have demonstrated that these negative impacts are not as severe as once thought. A recent 35-year long study, found no significant differences between parents of adult children with and without intellectual disabilities on measures of psychological well-being, depression, physical health, and divorce.

The aim for this study is therefore to evaluate the effectiveness of a culturally specific Psycho-social Training Intervention on disability on the knowledge and mental health of parents with intellectually disabled children, with an aim of rolling it out in Africa if it proves to be effective.

Research hypothesis:

The research hypothesis to be tested in this study is: The Psycho-social Training Intervention that will be developed will be more effective in improving psychological health for parents with intellectually disabled children than the usual health talk.

Methodology:

Research design: This study will use mixed methods design. An explanatory sequential design will be used. This is a design whereby qualitative data collection and analysis builds to quantitative data collection and analysis then finalizing with interpretation.

To complete the whole study, a phenomenological study using focus group discussions and indepth interviews will be followed by literature review and then a randomized trial will be done to test effectiveness of the developed intervention.

Section one: Qualitative part Design: The first part of this study will utilize phenomenological qualitative research design as it will focus on the lived experiences of Parents of Intellectually Disabled Children. A phenomenological design will help to understand the psychological issues encountered by Parents of Intellectually Disabled Children through their lived experiences. Details for this phase have been detailed in our qualitative paper.

Section two: Literature desk review and Design of the study's intervention:

Since this study will use a newly developed intervention, there is need to use participatory approaches, through focus group discussions with parents of intellectually disabled children in order to enhance acceptability and effectiveness of the intervention.

While some components of the psycho-social training intervention for this study will come from the findings in the qualitative study above, a systematic review of literature on similar interventions from elsewhere will be conducted to isolate aspects that will feed into the culturally relevant intervention to be developed for use in the third phase of the study. The third step, a desk review, will be done to contrast the current intervention from previous ones that have been developed for use in foreign countries by community staff.

The review of literature will follow this procedure:

Review dates and language: Literature to be reviewed will include those from the last ten years was searched, with mostly works in English language will be included in this review.

Databases: Databases to be searched for this purpose will include: Pubmed central, Hinari, and Google scholar. Grey literature, including thesis reports and another unpublished works will also be reviewed as well as engaging in personal contacts with seasoned authors in this field through emails and phone calls where possible. Hand searches and desk review of government websites for those countries that have done work in this area will also be undertaken to identify wider relevant literature.

Section three: Design of the intervention and piloting of the intervention:

The final stage in this phase will be the creation and then piloting of the intervention in order to assess the feasibility of intervention for use with parents who have intellectually disabled children, and to establish preliminary evidence of efficacy in reducing mental health problems among the parents. This will involve pretesting and modifying the intervention based on the pretesting results. The piloting will be done with 10 parents before the main study using clinic venues which will not be included in the main study.

Section four: Randomized Wait-list trial study:

The main study will be a randomized Waiting list-controlled trial. Children with intellectual disabilities, (as diagnosed by a psychologist or psychiatric clinical officer using a ten question questionnaire), will be consecutively referred and randomly allocated to the study in two sites. The intervention group will get Psycho-social Training Intervention while the waiting list (control) will continue getting the general health education that is done at disability clinics in the existing sites.

To avoid contamination, the intervention and the control will get their respective training on different days (Tuesdays-intervention groups session and Thursday-the control group sessions). The study will use blocked randomization (random permuted blocks) which is a common form of restricted randomization. This will ensure that subjects assigned to the experimental and waiting-control groups are balanced within blocks of, for example, five in one group and five in the other for every ten consecutively entered subjects. Follow-up, to check the impact of the intervention, will be done at six and twelve months from the time of intervention.

Study population: The study will recruit parents who are caring for intellectually disabled children using the inclusion criteria below.

Site and Sample Size and Sampling: The study will be conducted within catchment areas of two disability organizations that are operating in Mzuzu (St John of God), and Lilongwe (Children of Blessings Trust).

On sample size, three factors to be considered in the calculation of sample size are as follows: The level of statistical significance, normally 5%; The power, i.e. the probability to detect (reach statistical significance) for a given effect size, will be 90%; and The effect size is the difference between the two means you want to compare divided by the standard deviation. In this case, the affect size of 0.4 as found in recent meta-analysis for similar intervention, will be used for this calculation. This gives 81 participants per group. However, to factor in a 10% loss to follow-up, (8 subjects) will be added making the total number in each group to be 89.

Plan for data collection: A data collection questionnaire will be developed comprising questions on social-demographic data and associated variables in section one and questions based on "Self-Reported Questionnaire (SRQ)" to measure psychological distress in section two. Self-Reported Questionnaire has already been validated in Malawi. While Tumbuka is spoken in the rural northern region, many people in the city of Mzuzu speak Chichewa hence no problem is anticipated in participants understanding of the language. The entire questionnaire will be administered to all subjects in both groups at Baseline as well as at six and twelve months follow-up. These interviews will take 20 minutes each. The training will comprise of Ten- 40 minutes sessions conducted twice every week. Participant will be expected to attend all training sessions and transport to the venues will be reimbursed.

All research assistants who will be collecting data (under the supervision of the researcher) will be trained in the administration of the questionnaires and the methodology of the study.

The main study outcome: The main outcome measure will be psychological distress (Measured by Self-Reported Questionnaire.

Plan for data management and analysis Data for this study will be coded on a computer, cleaned and analyzed using Statistical package for social scientists.

At baseline and follow-up screening, the prevalence of common psychological health problems among carers will be calculated from the Self-Reported Questionnaire scores. Cases will be defined as those scoring 8 or above on the Self-Reported Questionnaire. Total number of cases, will be divided by total number of subjects to give the prevalence.

Since the outcome variables are categorical and continuous, Mann-Whitney test will be used to measure the impact of the intervention.

Plan for dissemination of results Findings of this study will be shared during Journal club sessions at the three clinic sites; Research Dissemination Conferences in Malawi and Sub-region; and manuscripts will be submitted for publication in peer reviewed journals.

Ethical Considerations:

Great care will be taken to ensure that all ethical to ensure that subjects are treated with respect allow for their right to refuse participation in the study, and conducting interviews in privacy. Further permission to carry out the study will be sought from the two institutional heads; ethical clearance will be sought from the College of medicine ethics committee; while written informed consent will be sought from all subjects before participating in the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included on the following criteria:

* Being carers of children with an intellectual disability, aged at least 18 years, for at least a year;
* Readiness to consent for the study on a voluntary basis, and
* Commitment to attend all training sessions, and
* Willingness to complete home assignments between training sessions.

Exclusion Criteria:

Subjects will be excluded on the following criteria:

* Aged less than 18 years,
* Having a psychiatric of being mentally unsound at the time of enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Psychological distress (Self reported Questionnaire {SRQ}) | 1 year
  SRQ screens for common psychological health problems using a 20 items scale

CONTACTS AND LOCATIONS:
Overall Officials: Don Mathanga, PhD, Study Chair — College of Medicine

IPD SHARING:
Plan to Share IPD: Yes
Yes

REFERENCES:
- [Background] Quinn, Mark, et al.